CLINICAL TRIAL: NCT02354599
Title: A Randomized, Single-center, Double-Blind, Placebo-Controlled Phase 1 Study to Evaluate Safety and Pharmacokinetics of Single Subcutaneous Injection of MT203 in Healthy Adult Japanese and Caucasian Male Participants
Brief Title: Single-Dose Study of MT203
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT203/CPH-001; U1111-1163-4003 (Registry Identifier: UTN (WHO)); JapicCTI-142699 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2014-11-07; First posted 2015-02-03 (Estimated); Results first posted 2016-06-20 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-05

CONDITIONS: Healthy Volunteers
Keywords: Randomized, double-blind, placebo-controlled, single-dose subcutaneous administration study
MeSH Terms: interventions — namilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- Cohort 1: MT203 80 mg (Experimental): Six Japanese participants will be randomized to receive a single dose of MT203 80 mg and 2 participants will be randomized to receive matched placebo subcutaneously.
  Interventions: Drug: MT203 80 mg or matching Placebo
- Cohort 1: MT203 80 mg matching placebo (Placebo Comparator): Six Japanese participants will be randomized to receive a single dose of MT203 80 mg and 2 participants will be randomized to receive matched placebo subcutaneously.
  Interventions: Drug: MT203 80 mg or matching Placebo
- Cohort 2: MT203 150 mg (Experimental): Six Japanese participants will be randomized to receive a single dose of MT203 150 mg and 2 participants will be randomized to receive matched placebo subcutaneously.
  Interventions: Drug: MT203 150mg or matching Placebo
- Cohort 2: MT203 150 mg matching placebo (Placebo Comparator): Six Caucasian participants will be randomized to receive a single dose of MT203 150 mg and 2 participants will be randomized to receive matched placebo subcutaneously.
  Interventions: Drug: MT203 150mg or matching Placebo
- Cohort 3: MT203 300 mg (Experimental): Six Japanese participants will be randomized to receive a single dose of MT203 300 mg and 2 participants will be randomized to receive matched placebo subcutaneously.
  Interventions: Drug: MT203 300 mg or matching placebo
- Cohort 3: MT203 300 mg matching placebo (Placebo Comparator): Six Japanese participants will be randomized to receive a single dose of MT203 300 mg and 2 participants will be randomized to receive matched placebo subcutaneously.
  Interventions: Drug: MT203 300 mg or matching placebo
- Cohort 4: MT203 150 mg (Experimental): Six Caucasian participants will be randomized to receive a single dose of MT203 150 mg and 2 participants will be randomized to receive matched placebo subcutaneously.
  Interventions: Drug: MT203 150mg or matching Placebo
- Cohort 4: MT203 150 mg matching placebo (Placebo Comparator): Six Caucasian participants will be randomized to receive a single dose of MT203 150 mg and 2 participants will be randomized to receive matched placebo subcutaneously
  Interventions: Drug: MT203 150mg or matching Placebo

INTERVENTIONS:
Drug: MT203 80 mg or matching Placebo — MT203 80 mg or matching placebo injection
  Other Names: Namilumab; Placebo
  Arms: Cohort 1: MT203 80 mg; Cohort 1: MT203 80 mg matching placebo
Drug: MT203 150mg or matching Placebo — MT203 150mg or matching placebo injection
  Other Names: Namilumab; Placebo
  Arms: Cohort 2: MT203 150 mg; Cohort 2: MT203 150 mg matching placebo; Cohort 4: MT203 150 mg; Cohort 4: MT203 150 mg matching placebo
Drug: MT203 300 mg or matching placebo — MT203 300 mg or matching placebo injection
  Other Names: Namilumab; Placebo
  Arms: Cohort 3: MT203 300 mg; Cohort 3: MT203 300 mg matching placebo

SUMMARY:
The purpose of this study is to evaluate safety, pharmacokinetics and pharmacodynamics of single subcutaneous injection of MT203 in healthy adult Japanese and Caucasian male participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called MT203 (Namilumab), which is a human immunoglobulin G1 (IgG1) mAb potently and specifically neutralizing human and macaque granulocyte macrophage colony stimulating factor (GM-CSF). This study will consist of Cohorts 1 to 3 for healthy Japanese participants and Cohort 4 for healthy Caucasian participants. Each cohort will be comprised of 8 participants, of whom 6 participants will be randomized to receive MT203 and 2 participants will be randomized to receive matched placebo.

The study population for the study will consist of 24 Japanese and 8 Caucasian healthy participants. Participants will be assigned to 4 cohorts which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need)::

Cohort 1:- MT203 80 mg (6 healthy Japanese participants); Matching Placebo (2 healthy Japanese participants) Cohort 2:- MT203 150 mg (6 healthy Japanese participants); Matching Placebo (2 healthy Japanese participants) Cohort 3:- MT203 300 mg (6 healthy Japanese participants); Matching Placebo (2 healthy Japanese participants) Cohort 4:- MT203 150 mg (6 healthy Caucasian participants); Matching Placebo (2 healthy Caucasian participants).

Dosing of the Caucasian participants (Cohort 4) may occur in parallel with dosing in Japanese participants (Cohorts 1 to 3). Dose escalation will occur in Japanese Cohorts, independent from Cohort 4. The dose escalation will only occur following a review of the blinded safety/tolerability data up to Day 15 from the previous cohort. All participants will receive a single dose on Day 1, admitted from Day -1 to Day 15. Participants will return to the study unit for the pharmacokinetic, pharmacodynamic and safety assessment on Days 22, 29, 43, 57, 71 and 85.

This trial will be conducted in Japan.Overall time to participate in this trial is 85 days.

ELIGIBILITY:
Inclusion Criteria: -

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant signs and dates a written, informed consent form and any required privacy authorizations prior to the initiation of any study procedures.
3. The participant is a healthy adult male of Japanese or Caucasian (born to Caucasian parents and grandparents).
4. The participant is aged 20 to 45 years, inclusive, at the time of informed consent.
5. The participant weighs at least 50 kilogram (kg) and has a body mass index (BMI) between 18.5 and 25.0 kilogram per square meter (kg/m2) (for Japanese) or between 18.5 and 30.0 kg/m2 (for Caucasian), inclusive at screening and Day-1.
6. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 18 weeks (126 days) after last dose.

Exclusion Criteria: -

1. The participant has received any investigational compound within 16 weeks (112 days) prior to the first dose of study medication.
2. The participant has received MT203 or other anti-granulocyte-macrophage colony stimulating factor (GM-CSF) drugs in a previous clinical study.
3. The participant has been vaccinated within 4 weeks (28 days) prior to the first dose of study medication or is scheduled to be vaccinated during the study.
4. The participant is an immediate family member, study site employee or may consent under duress.
5. The participant has uncontrolled, clinically significant neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, or endocrine disease or other abnormalities, which may impact the ability of the participant to participate or potentially confound the study results.
6. History of frequent or chronic infections or herpes zoster.
7. The participant has a history of or currently has significant pulmonary disease, inflammatory disease or autoimmune disease.
8. The participant has a known hypersensitivity to any component of the formulation of MT203.
9. The participant has a positive urine drug result for drugs of abuse at screening. 10. The participant has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 2 years prior to the screening visit or is unwilling to agree to abstain from alcohol and drugs throughout the study.

11. The participant has taken or requires excluded medications, supplements or food products listed in the Excluded Medications section throughout the study.

12. The participant intends to donate sperm during the course of this study or for 18 weeks after the last dose of study medication.

13. The participant has a history of cancer. 14. Presence, suspicion or history of active tuberculosis (TB) or latent TB infection.

15. The participant has a positive test result for hepatitis B virus (HBV) surface antigen (HBsAg), hepatitis B virus antibody (HBV surface virus antibody [HBsAb]/ HBV core antibody [HBcAb]), hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) antibody/antigen at screening. However, participants who are positive for HBsAb due to HBV vaccination are exempt.

16. The participant has used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum) within 4 weeks (28 days) prior to the first dose of study medication.

17. The participant has clinically relevant decreased lung function, example, forced expiratory volume in the first second (FEV1) less than (<) 70 percent (%) of the predicted value.

18. The participant has poor peripheral venous access. 19. The participant has undergone whole blood collection of at least 200 milliliter (mL) within 4 weeks (28 days) or at least 400 mL within 12 weeks (84 days) prior to the first dose of study medication.

20. The participant has undergone whole blood collection of at least 800 mL in total within 52 weeks (364 days) prior to the first dose of study medication.

21. The participant has undergone blood component collection within 2 weeks (14 days) prior to the start of study medication administration.

22. Participant has an abnormal (clinically significant) electrocardiogram (ECG) at screening or Day 1.

23. The participant has abnormal laboratory values at screening or Day-1 that suggest a clinically significant underlying disease or participant with the following laboratory abnormalities: Alanine transaminase (ALT) and/or aspartate transaminase (AST) greater than (>) 1.5 times the upper limit of normal or neutrophil counts and/or monocyte counts < the lower limit of normal.

24. Participant who, in the opinion of the investigator, is unlikely to comply with the protocol or is unsuitable for the study with any other reason.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Director, Study Director — Takeda
Locations (1):
- Kagoshima, Kagoshima-ken, Japan

REFERENCES:
- [Derived] Tanaka S, Harada S, Hiramatsu N, Nakaya R, Kawamura M. Randomized, double-blind, placebo-controlled, phase I study of the safety and pharmacokinetics of namilumab in healthy Japanese and Caucasian men . Int J Clin Pharmacol Ther. 2018 Nov;56(11):507-517. doi: 10.5414/CP203235. PMID 30168415

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant took part in the study at 1 investigative site in Japan from 25-November-2014 to 20-May-2015.
Pre-assignment Details: Healthy Japanese and Caucasian participants were enrolled in the study as 1 of the 4 cohorts Japanese participants in Cohort 1(MT203 80 milligram [mg]), Cohort 2 (MT203 150 mg), Cohort 3 (MT203 300 mg) and Caucasian participants in Cohort 4 (MT203 150 mg) to receive MT203, or matching placebo.
Groups:
- Cohort 1-3: Placebo: MT203 placebo -matching, injection, subcutaneously, once on Day 1 in the 15 days treatment period in Japanese participants.
- Cohort 1: MT203 80 mg: MT203 80 mg, injection, subcutaneously, once on Day 1 in the 15 days treatment period in Japanese participants.
- Cohort 2: MT203 150 mg: MT203 150 mg, injection, subcutaneously, once on Day 1 in the 15 days treatment period in Japanese participants.
- Cohort 3: MT203 300 mg: MT203 300 mg, injection, subcutaneously, once on Day 1 in the 15 days treatment period in Japanese participants.
- Cohort 4: Placebo: MT203 placebo-matching, injection, subcutaneously, once on Day 1 in the 15 days treatment period in Caucasian participants.
- Cohort 4: MT203 150 mg: MT203 150 mg, injection, subcutaneously, once on Day 1 in the 15 days treatment period in Caucasian participants.
Period: Overall Study
Arm/Group | Cohort 1-3: Placebo | Cohort 1: MT203 80 mg | Cohort 2: MT203 150 mg | Cohort 3: MT203 300 mg | Cohort 4: Placebo | Cohort 4: MT203 150 mg
Started | 6 | 6 | 6 | 6 | 2 | 6
Completed | 5 | 5 | 6 | 6 | 2 | 5
Not Completed | 1 | 1 | 0 | 0 | 0 | 1
Not completed — Pretreatment Event/Adverse Event | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAS) included all participants who received the study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1-3: Placebo | Cohort 1: MT203 80 mg | Cohort 2: MT203 150 mg | Cohort 3: MT203 300 mg | Cohort 4: Placebo | Cohort 4: MT203 150 mg | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 2 | 6 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.2 (8.89) | 26.0 (4.05) | 26.5 (7.79) | 24.2 (6.85) | 28.0 (7.07) | 36.0 (6.29) | 28.2 (7.56)
Sex/Gender, Customized [Number; unit: participants]
  Male | 6 | 6 | 6 | 6 | 2 | 6 | 32
Smoking Classification [Number; unit: participants]
  Never Smoked | 4 | 3 | 5 | 2 | 2 | 5 | 21
  Ex-smoker | 2 | 3 | 1 | 4 | 0 | 1 | 11
Alcohol Classification [Number; unit: participants]
  Drank a few days per week | 2 | 0 | 1 | 1 | 0 | 2 | 6
  Drank a few days per month | 0 | 2 | 3 | 3 | 2 | 2 | 12
  Never drank | 4 | 4 | 2 | 2 | 0 | 2 | 14
Caffeine Classification [Number; unit: participants]
  Had caffeine consumption | 2 | 3 | 1 | 2 | 2 | 3 | 13
  Had no caffeine consumption | 4 | 3 | 5 | 4 | 0 | 3 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAE)
Time Frame: Baseline up to Day 85
Population: The safety analysis set was defined as all participants who received the study medication.
Measure: Number; unit: participants
Arm/Group | Cohort 1-3: Placebo | Cohort 1: MT203 80 mg | Cohort 2: MT203 150 mg | Cohort 3: MT203 300 mg | Cohort 4: Placebo | Cohort 4: MT203 150 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 2 | 6
participants | 3 | 3 | 1 | 1 | 1 | 5

2. Primary Outcome: Number of Participants With TEAEs Related to Vital Signs
Time Frame: Baseline up to Day 85
Population: The safety analysis set was defined as all participants who received the study medication.
Measure: Number; unit: participants
Arm/Group | Cohort 1-3: Placebo | Cohort 1: MT203 80 mg | Cohort 2: MT203 150 mg | Cohort 3: MT203 300 mg | Cohort 4: Placebo | Cohort 4: MT203 150 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 2 | 6
participants | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With TEAEs Related to Body Weight
Time Frame: Baseline up to Day 85
Population: The safety analysis set was defined as all participants who received the study medication.
Measure: Number; unit: participants
Arm/Group | Cohort 1-3: Placebo | Cohort 1: MT203 80 mg | Cohort 2: MT203 150 mg | Cohort 3: MT203 300 mg | Cohort 4: Placebo | Cohort 4: MT203 150 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 2 | 6
participants | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With TEAEs Related to 12-lead Electrocardiograms (ECG)
Time Frame: Baseline up to Day 85
Population: The safety analysis set was defined as all participants who received the study medication.
Measure: Number; unit: participants
Arm/Group | Cohort 1-3: Placebo | Cohort 1: MT203 80 mg | Cohort 2: MT203 150 mg | Cohort 3: MT203 300 mg | Cohort 4: Placebo | Cohort 4: MT203 150 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 2 | 6
participants | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With TEAEs Related to Lung Functioning Monitoring
Time Frame: Baseline up to Day 85
Population: The safety analysis set was defined as all participants who received the study medication.
Measure: Number; unit: participants
Arm/Group | Cohort 1-3: Placebo | Cohort 1: MT203 80 mg | Cohort 2: MT203 150 mg | Cohort 3: MT203 300 mg | Cohort 4: Placebo | Cohort 4: MT203 150 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 2 | 6
participants | 0 | 1 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With TEAEs Related to Hematology, Serum Chemistry and Urinalysis
Time Frame: Baseline up to Day 85
Population: The safety analysis set was defined as all participants who received the study medication.
Measure: Number; unit: participants
Arm/Group | Cohort 1-3: Placebo | Cohort 1: MT203 80 mg | Cohort 2: MT203 150 mg | Cohort 3: MT203 300 mg | Cohort 4: Placebo | Cohort 4: MT203 150 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 2 | 6
participants
  Hematology | 0 | 0 | 0 | 0 | 0 | 0
  Serum Chemistry | 0 | 0 | 0 | 0 | 0 | 0
  Urinalysis | 1 | 1 | 0 | 1 | 1 | 0

7. Secondary Outcome: Area Under the Serum Concentration-Time Curve From Time 0 to Infinity (AUC(0-inf)) of MT203
Time Frame: Predose and at multiple time points (up to 84 days) post-dose
Population: The pharmacokinetic analysis set as defined as all participants who received the study medication without any major protocol deviations, and met the minimum procedure specified in the study protocol and had evaluable pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: nanogram*day per milliliter (ng*day/mL)
Arm/Group | Cohort 1: MT203 80 mg | Cohort 2: MT203 150 mg | Cohort 3: MT203 300 mg | Cohort 4: MT203 150 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
nanogram*day per milliliter (ng*day/mL) | 315573.3 (47464.44) | 575180.7 (126751.71) | 1238496.3 (222651.06) | 559689.3 (188835.67)

8. Secondary Outcome: Area Under the Serum Concentration-Time Curve From Time 0 to Time 84 Days (AUC(0-84d)) of MT203
Time Frame: Predose and at multiple time points (up to 84 days) post-dose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng*day/mL
Arm/Group | Cohort 1: MT203 80 mg | Cohort 2: MT203 150 mg | Cohort 3: MT203 300 mg | Cohort 4: MT203 150 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng*day/mL | 286383.2 (44732.15) | 502017.5 (116382.43) | 1106605.2 (207794.23) | 451596.7 (133571.47)

9. Secondary Outcome: Maximum Observed Serum Concentrations (Cmax) of MT203
Time Frame: Predose and at multiple time points (up to Day 84) post-dose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Cohort 1: MT203 80 mg | Cohort 2: MT203 150 mg | Cohort 3: MT203 300 mg | Cohort 4: MT203 150 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
nanogram per milliliter (ng/mL) | 8381.3 (1848.65) | 15354.5 (5097.64) | 32580.7 (9061.85) | 10826.7 (3220.93)

10. Secondary Outcome: Terminal Elimination Half-Life (T1/2) of MT203
Time Frame: Predose and at multiple time points (up to 84 days) post-dose
Population: as for outcome 7
Measure: Median (Full Range); unit: day
Arm/Group | Cohort 1: MT203 80 mg | Cohort 2: MT203 150 mg | Cohort 3: MT203 300 mg | Cohort 4: MT203 150 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
day | 23.75 [22.3 to 25.7] | 26.20 [22.6 to 43.0] | 26.15 [22.7 to 31.1] | 32.60 [25.2 to 44.9]

11. Secondary Outcome: Plasma Total Granulocyte-Macrophage Colony Stimulating Factor (GM-CSF) Concentration
Time Frame: Baseline, Hour 24, 72, 120, 168, 240, 336 hours, Day 21, 28, 42, 56, 70, 84
Population: The pharmacodynamic analysis set was defined as all participants who received the study medication without any major protocol deviations, and met the minimum procedure specified in the study protocol and had evaluable pharmacodynamic data.
Measure: Mean (Standard Deviation); unit: picogram per milliliter (pg/mL)
Arm/Group | Cohort 1: MT203 80 mg | Cohort 2: MT203 150 mg | Cohort 3: MT203 300 mg | Cohort 4: MT203 150 mg | Cohort 1-3: Placebo | Cohort 4: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 2
picogram per milliliter (pg/mL)
  Baseline | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  24 Hours | 0.000 (0.0000) | 0.000 (0.0000) | 9.123 (22.3475) | 14.857 (23.0308) | 0.000 (0.0000) | 0.000 (0.0000)
  72 Hours | 123.535 (20.4004) | 131.165 (25.2255) | 155.707 (37.5200) | 134.788 (39.9181) | 0.000 (0.0000) | 0.000 (0.0000)
  120 Hours | 215.698 (33.8697) | 233.063 (46.0860) | 277.878 (57.0774) | 248.055 (79.1963) | 0.000 (0.0000) | 0.000 (0.0000)
  168 Hours | 291.852 (48.4269) | 314.218 (65.0007) | 375.772 (72.3014) | 361.720 (113.4442) | 0.000 (0.0000) | 0.000 (0.0000)
  240 Hours | 387.628 (60.4318) | 415.098 (88.4198) | 489.127 (72.4588) | 493.835 (113.3446) | 0.000 (0.0000) | 0.000 (0.0000)
  336 Hours | 483.353 (77.2963) | 554.973 (122.5254) | 675.010 (96.1891) | 565.527 (137.2089) | 0.000 (0.0000) | 0.000 (0.0000)
  21 Days | 733.440 (330.8767) | 710.998 (202.6718) | 859.977 (160.9109) | 677.693 (194.5259) | 0.000 (0.0000) | 0.000 (0.0000)
  28 Days | 653.467 (111.0059) | 758.195 (157.6988) | 951.438 (207.3810) | 781.040 (167.7037) | 0.000 (0.0000) | 0.000 (0.0000)
  42 Days | 547.093 (81.0675) | 740.245 (245.6498) | 807.632 (193.1090) | 828.695 (271.3573) | 0.000 (0.0000) | 0.000 (0.0000)
  56 Days | 431.300 (94.4867) | 633.093 (186.5863) | 758.747 (238.7338) | 617.653 (192.0337) | 0.000 (0.0000) | 0.000 (0.0000)
  70 Days | 325.750 (67.8796) | 440.092 (126.7378) | 668.387 (181.7359) | 467.965 (173.5354) | 0.000 (0.0000) | 0.000 (0.0000)
  84 Days | 240.712 (44.5704) | 366.078 (200.2973) | 545.100 (151.8562) | 379.647 (189.7192) | 0.000 (0.0000) | 0.000 (0.0000)

12. Secondary Outcome: Number of Participants With Positive Response for Anti MT203 Antibody
Time Frame: Baseline, Hour 168, 336, Day 42, 84
Population: The safety analysis set was defined as all participants who received the study medication.
Measure: Number; unit: participants
Arm/Group | Cohort 1: MT203 80 mg | Cohort 2: MT203 150 mg | Cohort 3: MT203 300 mg | Cohort 4: MT203 150 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
participants
  Baseline | 0 | 0 | 0 | 0
  168 Hours | 0 | 1 | 1 | 2
  336 Hours | 1 | 1 | 0 | 1
  42 Days | 0 | 2 | 0 | 1
  84 Days | 0 | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug on Day 1 up to Day 85
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Cohort 1-3: Placebo | Cohort 1: MT203 80 mg | Cohort 2: MT203 150 mg | Cohort 3: MT203 300 mg | Cohort 4: Placebo | Cohort 4: MT203 150 mg
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/2 | 1/6
Other Adverse Events (participants affected / at risk) | 3/6 | 3/6 | 1/6 | 1/6 | 1/2 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1-3: Placebo (N=6) | Cohort 1: MT203 80 mg (N=6) | Cohort 2: MT203 150 mg (N=6) | Cohort 3: MT203 300 mg (N=6) | Cohort 4: Placebo (N=2) | Cohort 4: MT203 150 mg (N=6)
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1-3: Placebo (N=6) | Cohort 1: MT203 80 mg (N=6) | Cohort 2: MT203 150 mg (N=6) | Cohort 3: MT203 300 mg (N=6) | Cohort 4: Placebo (N=2) | Cohort 4: MT203 150 mg (N=6)
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Blood urine present (Investigations) | 1 | 1 | 0 | 0 | 1 | 0
Forced vital capacity decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Protein urine present (Investigations) | 0 | 1 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.